CLINICAL TRIAL: NCT00662220
Title: High-dose Versus Standard-dose Weight-based Ribavirin in Combination With Peginterferon Alfa-2a for Patients Infected With Hepatitis C Virus Genotype 1 or 4
Brief Title: High-dose Ribavirin in Treatment of Chronic Hepatitis C Genotype 1 or 4
Acronym: VIRID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the arrival of DAAs replacing standard of care for genotype 1 patients the VIRID study had to be terminated.
Sponsor: Foundation for Liver Research (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV07-01; 2007-005344-25 (EudraCT Number)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Hepatitis C
Keywords: chronic; hepatitis C; ribavirin; SVR; genotype one; genotype four
MeSH Terms: conditions — Hepatitis C, Chronic; Bronchiolitis Obliterans Syndrome; Hepatitis C | interventions — Ribavirin; peginterferon alfa-2a; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dose (Active Comparator): Standard-dose ribavirin (12-15 mg/kg/day) in combination with peginterferon 180µg QW
  Interventions: Drug: ribavirin
- High dose (Experimental): High-dose ribavirin (25-29 mg/kg/day) in combination with peginterferon 180µg QW
  Interventions: Drug: ribavirin

INTERVENTIONS:
Drug: ribavirin — 25-29 mg/kg/day
  Other Names: Copegus; Pegasys; NeoRecormon
  Arms: High dose
Drug: ribavirin — 12-15 mg/kg/day
  Other Names: Copegus; Pegasys; NeoRecormon
  Arms: Standard dose

SUMMARY:
Optimal ribavirin dosages are essential in achieving SVR (sustained virological response). Several studies have shown higher SVR rates in patients receiving higher doses of ribavirin. Therefore we propose a randomized controlled open label multicenter trial to investigate wether high (25-29mg/kg) dose ribavirin can improve outcome in patients in infected with hepatitis C virus genotype 1 or 4 compared to standard dose (12-15mg/kg).

DETAILED DESCRIPTION:
Optimal ribavirin dosages are essential in achieving SVR. The initial evidence supporting higher doses of ribavirin for peginterferon alfa-2b comes from a secondary analysis of the pivotal multicenter trial of peginterferon alfa-2b and ribavirin. Patients receiving more than 10.6 mg/kg/day ribavirin experienced significantly higher SVR rates (48% vs. 38%). A large multicenter trial designed to test standard dose ribavirin (1000-1200 mg/day) versus low-dose ribavirin (800 mg/day) in combination with peginterferon alfa-2a, showed 52% SVR in the standard dose group versus 41% in the low-dose group for genotype 1 infected patients. In the pooled data from two pivotal studies with peginterferon alfa-2a and ribavirin, the probability of achieving an SVR for genotype 1 patients was influenced by the ribavirin dose per kg body weight. A 40-50% increase in the probability of SVR was found for a 12-16 mg/kg dose increase of ribavirin. For peginterferon alfa-2b it was also shown among genotype 1 patients, that weight-based ribavirin (800-1400 mg/day) leads to higher SVR rates compared to fixed dose ribavirin (800 mg/day) (34% vs. 29%). Moreover, ribavirin dosing up to 1400 mg/day was safe and the rate of treatment discontinuation was the same for both treatment groups. In a small pilot study, 10 genotype 1 patients with a high baseline load were treated with peginterferon alfa-2a and individualized high-dose ribavirin in order to achieve a ribavirin target concentration in serum of 15 μmol/l. The mean ribavirin dose of 2540 mg/day (range 1600-3600 mg/day) was high, but resulted in 90% SVR. All patients experienced severe anemia, which was treated with concomitant epoetin beta and blood transfusion.

As mentioned before, the main concern of high-dose ribavirin will be a dose-dependent hemolytic anemia and the addition of epoetin alfa has shown significant increase of haemoglobin during (peg)interferon/ribavirin therapy. Erythropoietin doses from 9,000 to 60,000 IU/week have been used in order keep the highest possible ribavirin doses. A recent trial showed a significant higher SVR rate in genotype 1 patients treated with peginterferon alfa-2b, increased dose ribavirin (15.2 mg/kg/day) and epoetin alfa than in patients treated with peginterferon alfa-2b and standard dose ribavirin (13.3 mg/kg/day) with or without epoetin alfa. Using the standard ribavirin dose, routine use of erythropoietin significantly decreased the frequency of anemia and the mean ribavirin dose reduction. Moreover, with the addition of erythropoietin, a significant higher mean dose could be given to patients in the increased ribavirin dose arm.

ELIGIBILITY:
Inclusion Criteria:

* hepatitis C genotype 1 or 4
* high viral load (>400000 IU/ml)
* indication for antiviral treatment or patient's desire for antiviral treatment
* hepatitis C treatment naive
* liver biopsy within 3 years of screening visit or when biopsy is contraindicated e.g in patients with clotting diseases or when a patient refuses to undergo a new biopsy in case the liver biopsy is older than 3 years, substitution by fibroscan is allowed.
* age 18-70 years

Exclusion Criteria:

* serum bilirubin >35 μmol/l
* albumin <36 g/l
* prothrombin time >4 sec prolonged
* platelets <90x109/l
* decompensated cirrhosis (Child-Pugh Grade B or C)
* hepatic imaging (ultrasound, CT or MRI) with the evidence of hepatocellular carcinoma (hepatic imaging should be performed within 3 months prior to screening for cirrhotic patients and within 6 months prior to screening for non-cirrhotic patients)
* alcoholic liver disease (indicator: MCV>100)
* obesity induced liver disease (indicators: steatosis proven by biopsy or ultrasound in association with a body mass index >30)
* drug related liver disease (indicator: positive history of hepatic toxic drug intake with a causal relation)
* auto-immune hepatitis (indicators: IgG >30g/l, anti smooth-muscle or antinuclear antibodies titer ³1:40)
* hemochromatosis (indicator: ferritin >1000 μg/l)
* Wilson's disease (indicator: ceruloplasmin (<0.2 g/l)
* alpha-1 antitrypsin deficiency (indicator alpha-1 antitrypsin <0.8 g/L)
* co-infection with hepatitis B virus or human immunodeficiency virus (HIV)
* any cardiovascular dysfunction (e.g. cardiac decompensation, myocardial infarction, present or history of arrythmia)
* other medical illness that might interfere with this study: significant pulmonary or renal dysfunction, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g.: steroid therapy, organ transplants other than cornea and hair transplant)
* contra-indications for peginterferon and/or ribavirin:
* severe psychiatric disorder, such as major psychoses, suicidal ideation, suicidal attempt and/or manifest depression. Severe depression would include the following: (a) subjects who have been hospitalized for depression, (b) subjects who have received electroconvulsive therapy for depression, or (c) subjects whose depression has resulted in a prolonged absence of work and/or significant disruption of daily functions. Subjects with a history of mild depression may be considered for entry into the protocol provided that a pretreatment assessment of the subject's mental status supports that the subject is clinically stable and that there is ongoing evaluation of the patient's mental status during the study
* visual symptoms related to retinal abnormalities
* pregnancy, breast-feeding or inadequate contraception
* thalassemia, spherocytosis
* females who are pregnant or intending to become pregnant or male partners of females who are pregnant or intending to become pregnant
* absolute neutrophil count (ANC) <1.40x109/l
* hemoglobin (Hb) <7.5 mmol/l (female) or <8.1 mmol/l (male)
* serum creatinine concentration >1.5 times the upper limit of normal at screening
* substance abuse, such as I.V. drugs or alcohol (indicator: >28 drinks/week). If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 1 year
* any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-04; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
HCV-RNA negativity by qualitative assay 24 weeks after end of treatment (sustained virological response, SVR) | 72 weeks

SECONDARY OUTCOMES:
HCV-RNA negativity at week 4 (rapid virological response, RVR) | 4 weeks
HCV-RNA negativity at week 12 (complete early virological response, cEVR) | 12 weeks
HCV-RNA ≥ 2log10 drop at week 12, but HCV-RNA still detectable (partial early virological response, pEVR) | 12 weeks
HCV- RNA negativity at week 48 (end of treatment response, ETR) | 48 weeks
Relapse rate after ETR | 48 weeks - end of follow up
Safety and tolerability of high-dose daily ribavirin (serious adverse events, grade 4 NCI toxicity, percentage of patients completing treatment on full or >80% of total intended dose and reasons for dose adjustments) | week 0 till end of follow up
Biochemical response (normalization of serum ALT at the end of therapy and at the end of follow-up) | week 0 - end of follow up
Health related quality of life and psychopathology before, during and after treatment by SF-36 and SCL-90 questionnaires | week 0 - week 72

CONTACTS AND LOCATIONS:
Overall Officials: R J de Knegt, MD PhD, Principal Investigator — Erasmus Medical Center; J PH Drenth, MD PhD, Principal Investigator — St Radboud Medical Center
Locations (27):
- Netherlands (27):
  - Rijnstate, Arnhem, Gelderland
  - St. Radboud University Medical Center, Nijmegen, Gelderland
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Atrium Medisch Centrum, Heerlen, Limburg
  - Amphia hospital, Breda, North Brabant
  - Catharina hospital, Eindhoven, North Brabant
  - Twee Steden hospital, Tilburg, North Brabant
  - St. Elisabeth hospital, Tilburg, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Slotervaart hospital, Amsterdam, North Holland
  - VU Medisch Centrum, Amsterdam, North Holland
  - Onze Lieve Vrouwen Gasthuis, Amsterdam, North Holland
  - Spaarne Ziekenhuis, Hoofddorp, North Holland
  - Deventer hospital, Deventer, Overijssel
  - Groningen University Medical Center, Groningen, Provincie Groningen
  - St. Lucas hospital, Winschoten, Provincie Groningen
  - IJsselland hospital, Capelle aan den IJssel, South Holland
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Albert Schweitzer hospital, Dordrecht, South Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - St Franciscus hospital, Rotterdam, South Holland
  - Erasmus MC University Medical Center, Rotterdam, South Holland
  - Maasstad hospital, Rotterdam, South Holland
  - HAGA Ziekenhuis, The Hague, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht, Utrecht
  - Walcheren hospital, Flushing, Zeeland
  - ZorgSaam Hospital, Terneuzen, Zeeland

REFERENCES:
- See also: Study website — http://www.virid.nl